CLINICAL TRIAL: NCT03207009
Title: A Phase 3 Single Arm Study Evaluating the Efficacy and Safety of Gene Therapy in Subjects With Transfusion-dependent β-Thalassemia by Transplantation of Autologous CD34+ Stem Cells Transduced Ex Vivo With a Lentiviral βA-T87Q-Globin Vector in Subjects ≤50 Years of Age
Brief Title: A Study Evaluating the Efficacy and Safety of the LentiGlobin® BB305 Drug Product in Participants With Transfusion-Dependent β-Thalassemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGB-212
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — betibeglogene autotemcel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LentiGlobin BB305 Drug Product (Experimental): LentiGlobin BB305 Drug Product (autologous CD34+ cell-enriched population that contains cells transduced with LentiGlobin BB305 lentiviral vector encoding human βA-T87Q-globin)
  Interventions: Genetic: LentiGlobin BB305 Drug Product

INTERVENTIONS:
Genetic: LentiGlobin BB305 Drug Product — LentiGlobin BB305 Drug Product is administered by IV infusion following myeloablative conditioning with busulfan.
  Other Names: betibeglogene autotemcel

SUMMARY:
This is a single-arm, multi-site, single-dose, Phase 3 study in approximately 18 participants less than or equal to (<=) 50 years of age with transfusion-dependent β-thalassemia (TDT), who have a β0/β0, β0/IVS-I-110, or IVS-I-110/IVS-I-110 genotype. The study will evaluate the efficacy and safety of autologous hematopoietic stem cell transplantation (HSCT) using LentiGlobin BB305 Drug Product.

ELIGIBILITY:
Inclusion Criteria:

• Participants less than or equal to (<=) 50 years of age at the time of consent or assent (as applicable), and able to provide written consent (adults, or legal guardians, as applicable) or assent (adolescents or children). Provided that the data monitoring committee (DMC) has approved enrolling participants younger than 5 years of age, participants younger than 5 years of age may be enrolled if they weigh a minimum of 6 kilograms (kg) and are reasonably anticipated to be able to provide at least the minimum number of cells required to initiate the manufacturing process.

* Diagnosis of TDT with a history of at least 100 milliliter per kilogram per year (mL/kg/year) of pRBCs in the 2 years preceding enrollment (all participants), or be managed under standard thalassemia guidelines with >= 8 transfusions of pRBCs per year in the 2 years preceding enrollment (participants >=12 years).
* Clinically stable and eligible to undergo HSCT.
* Treated and followed for at least the past 2 years in a specialized center that maintained detailed medical records, including transfusion history.

Exclusion Criteria:

* Presence of a mutation characterized as other then β0 (e.g., β+, βE, βC) on at least one β-globin gene (HBB) allele.
* Positive for presence of human immunodeficiency virus type 1 or 2 (HIV-1 and HIV-2), hepatitis B virus (HBV), or hepatitis C (HCV).
* A white blood cell (WBC) count less than (<) 3×10^9/liter (L), and/or platelet count <100×10^9/L not related to hypersplenism.
* Uncorrected bleeding disorder.
* Any prior or current malignancy.
* Prior HSCT.
* Advanced liver disease.
* A cardiac T2* <10 ms by MRI.
* Any other evidence of severe iron overload that, in the investigator's opinion, warrants exclusion.
* Participation in another clinical study with an investigational drug within 30 days of Screening.
* Any other condition that would render the participant ineligible for HSCT, as determined by the attending transplant physician or investigator.
* Prior receipt of gene therapy.
* Pregnancy or breastfeeding in a postpartum female or absence of adequate contraception for fertile participant.
* A known and available human leukocyte antigen (HLA) matched family donor.
* Any contraindications to the use of granulocyte colony stimulating factor (G-CSF) and plerixafor during the mobilization of hematopoietic stem cells and any contraindications to the use of busulfan and any other medicinal products required during the myeloablative conditioning, including hypersensitivity to the active substances or to any of the excipients.

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Himal L Thakar, MD, Study Director — Genetix Biotherapeutics Inc.
Locations (9):
- United States (3):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hopital d'enfants de la Timone, Marseille, France
- Germany (2):
  - Hannover Medical School, Hanover
  - University of Heidelberg, Heidelberg
- General Hospital of Thessaloniki 'G.Papanikolaou', Thessaloniki, Greece
- IRCCS Ospedale Pediatrico Babino Gesu, Rome, Italy
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Bluebird bio is committed to transparency. Appropriately de-identified patient-level datasets and supporting documents may be shared (if contractually or otherwise legally permitted) following completion of this study, submission of all applicable regulatory submissions and consistent with criteria established by bluebird bio and/or industry best practices to protect confidential information and maintain the privacy of study participants. For enquiries, please contact us at datasharing@bluebirdbio.com.

REFERENCES:
- [Derived] Kwiatkowski JL, Walters MC, Hongeng S, Yannaki E, Kulozik AE, Kunz JB, Sauer MG, Thrasher AJ, Thuret I, Lal A, Tao G, Ali S, Thakar HL, Elliot H, Lodaya A, Lee J, Colvin RA, Locatelli F, Thompson AA. Betibeglogene autotemcel gene therapy in patients with transfusion-dependent, severe genotype beta-thalassaemia (HGB-212): a non-randomised, multicentre, single-arm, open-label, single-dose, phase 3 trial. Lancet. 2024 Nov 30;404(10468):2175-2186. doi: 10.1016/S0140-6736(24)01884-1. Epub 2024 Nov 8. PMID 39527960

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 study centers in France, Germany, Greece, Italy, United Kingdom, and United States, of which 8 active centers had enrolled participants from 08 June 2017 to 15 November 2022.
Pre-assignment Details: A total of 19 participants were enrolled, of which 18 participants aged <=50 years were treated with LentiGlobin BB305 Drug Product.
Groups:
- LentiGlobin BB305 Drug Product: Participants <=50 years of age received a single intravenous (IV) infusion of LentiGlobin BB305 Drug Product at a dose of >=5.0 × 10^6 CD34+ cells/kilogram (kg) body weight on Day 1 after myeloablative conditioning with busulfan (4 days of conditioning followed by at least 48 hours of washout) (termed the Transplant population).
Period: Overall Study
Arm/Group | LentiGlobin BB305 Drug Product
Started | 19
Intent-to-Treat (ITT) Population (ITT population included all 19 participants who initiated any study procedures, beginning with mobilization by G-CSF and/or plerixafor.) | 19
Transplant Population (TP) (TP included all participants who received beti-cel.) | 18
Completed | 18
Not Completed | 1
Not completed — Withdrew consent prior to conditioning | 1

BASELINE CHARACTERISTICS:
Population: Data are analyzed at times based on ITT population which included all 19 participants who initiated any study procedures, beginning with mobilization by G-CSF and/or plerixafor.
Groups:
- LentiGlobin BB305 Drug Product: Participants <=50 years of age received a single IV infusion of LentiGlobin BB305 Drug Product at a dose of >=5.0 × 10^6 CD34+ cells/kg body weight on Day 1 after myeloablative conditioning with busulfan (4 days of conditioning followed by at least 48 hours of washout) (termed the Transplant population).
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have Achieved Transfusion Independence (TI)
Description: TI was defined as a weighted average hemoglobin (Hb) >= 9 grams per deciliter (g/dL) without any packed red blood cell (pRBC) transfusions for a continuous period of >= 12 months at any time during the study after drug product infusion.
Time Frame: From 12 to 24 months post-transplant
Population: TP included all participants who received beti-cel. Participant evaluable for TI are defined as participant who have achieved TI, have not achieved TI in their parent study, or completed their parent study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
Percentage of participants | 88.9 [65.3 to 98.6]

2. Secondary Outcome: Percentage of Participants Who Have Achieved Transfusion Independence (TI) at Month 24
Description: as for outcome 1
Time Frame: At Month 24 post-transplant
Population: TP included all participants who received beti-cel. Participants evaluable for TI are defined as participants who have achieved TI, have not achieved TI in their parent study, or completed their parent study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
Percentage of participants | 88.9 [65.3 to 98.6]

3. Secondary Outcome: Duration of Transfusion Independence (TI)
Description: Duration of TI was calculated as the time from the start of TI (i.e. first Hb >=9 with no transfusions in the preceding 60 days) up to the last available Hb at which the TI criteria are still met using Kaplan-Meier methodology.
Time Frame: From start of TI up to Month 24 (actual maximum time frame of up to approximately 25 months due to visit window)
Population: TP included all participants who received beti-cel. Participants evaluable for TI are defined as participants who have achieved TI, have not achieved TI in their parent study, or completed their parent study. Here, "overall number of participants analyzed" signifies those participants who achieved TI. Data are presented through the Month 24 Visit based on calendar dates and including visit windows.
Measure: Median (Full Range); unit: Months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 16
Months | 20.86 [13.1 to 25.4]

4. Secondary Outcome: Time From Drug Product Infusion to Achievement of Transfusion Independence (TI)
Description: Time from drug product infusion to achievement of TI was calculated as the time from drug product infusion to the first hemoglobin at which a participant can be declared as TI (that is to 'start of TI + >= 12 months', dependent on Hb lab schedule).
Time Frame: From drug product infusion to start of TI (up to Month 24 [actual maximum time frame of up to approximately 25 months due to visit window])
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 16
Months | 15.67 [14.8 to 24.5]

5. Secondary Outcome: Weighted Average Hemoglobin (Hb) During Transfusion Independence (TI)
Description: Weighted average Hb was defined as the weighted average of Hb values without any pRBC transfusions in the proceeding 60 days for a given subject. Ratio of the time between two Hb values and the time between the first and the last Hb values was used as the weight for calculation.
Time Frame: Timeframe varied by subject. For a given subject, the endpoint was calculated from 60 days after the last pRBC transfusion (so transfused blood did not confound the weighted average calculation) through the Month 24 Visit for that subject.
Population: TP included all participants who received beti-cel. Participants evaluable for TI are defined as participants who have achieved TI, have not achieved TI in their parent study, or completed their parent study. Here, "overall number of participants analyzed" signifies those participants who achieved TI.
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 16
gram per deciliter (g/dL) | 10.817 (1.2535)

6. Secondary Outcome: Percentage of Participants Who Meet the Definition of Transfusion Reduction (TR)
Description: TR was defined as demonstration of a 60 percent (%) reduction in the annualized volume of pRBC transfusion requirements (in milliliter per kilogram [mL/kg]) in the post-treatment time period from 12 Months post-drug product infusion through Month 24 compared to the annualized mL/kg pRBC transfusion requirement during the 24 months prior to study enrollment.
Time Frame: From 12 to 24 months post-transplant
Population: TP included all participants who received beti-cel. Participants evaluable for TI are defined as participants who have achieved TI, have not achieved TI in their parent study, or completed their parent study. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
Percentage of participants | 94.4 [72.7 to 99.9]

7. Secondary Outcome: Percentage of Participants Who Had a Reduction of At Least 50%, 60%, 75%, 90% or 100% in the Annualized pRBCs Transfusion Volume
Description: Percentage of participants with a reduction in the annualized mL/kg pRBCs transfused from 12 months post-drug product infusion through Month 24 (approximately a 12-month period) of at least 50%, 60%, 75%, 90% or 100% compared to the annualized mL/kg pRBC transfusion requirement during the 24 months prior to enrollment.
Time Frame: 12 months post-drug product infusion through Month 24
Population: TP included all participants who received beti-cel.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
Percentage of participants
  Reduction at >= 50% | 94.4 [72.7 to 99.9]
  Reduction at >= 60% | 94.4 [72.7 to 99.9]
  Reduction at >= 75% | 94.4 [72.7 to 99.9]
  Reduction at >= 90% | 94.4 [72.7 to 99.9]
  Reduction at 100% | 88.9 [65.3 to 98.6]

8. Secondary Outcome: Annualized Number of pRBC Transfusions
Description: Annualized number of pRBC transfusions from 12 months post-drug product infusion through Month 24 was reported.
Time Frame: From 12 months post-drug product infusion through Month 24
Population: TP included all participants who received beti-cel.
Measure: Mean (Standard Deviation); unit: pRBC transfusions per year
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
pRBC transfusions per year | 0.68 (2.701)

9. Secondary Outcome: Annualized Volume of pRBC Transfusions
Description: Annualized volume of pRBC transfusions from 12 months post-drug product infusion through Month 24 compared to the annualized volume of transfusions during the 24 months prior to enrollment.
Time Frame: From 12 to 24 months post-transplant
Population: TP included all participants who received beti-cel.
Measure: Mean (Standard Deviation); unit: milliliter/kilogram/year (mL/kg/year)
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
milliliter/kilogram/year (mL/kg/year) | 11.589 (47.4080)

10. Secondary Outcome: Time From Drug Product Infusion to Last pRBC Transfusion
Description: Time from drug product infusion to last pRBC transfusion was reported.
Time Frame: From start of drug product infusion up to Month 24
Population: TP included all participants who received beti-cel.
Measure: Median (Full Range); unit: months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
months | 0.986 [0.00 to 23.36]

11. Secondary Outcome: Time From Last pRBC Transfusion to 24 Months
Description: Time From Last pRBC Transfusion to the Month 24 was reported.
Time Frame: From last pRBC Transfusion up to Month 24 (actual maximum time frame of up to approximately 27 months due to visit window)
Population: TP included all participants who received beti-cel. Data are presented through the Month 24 Visit based on calendar dates and including visit windows.
Measure: Median (Full Range); unit: Months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
Months | 23.211 [0.16 to 27.47]

12. Secondary Outcome: Weighted Average Nadir Hemoglobin (Hb)
Description: The weighted average nadir Hb was defined as the most recent Hb prior to each pRBC transfusion, on the day of transfusion or within 3 days and, if there was a period of more than 60 days without transfusion, all Hb records between Day 61 and last follow-up or next transfusion (inclusive) was included. The weighted average nadir Hb during the period of 12 months post-drug product infusion to Month 24 was compared to the weighted average nadir Hb during the 24 months prior to enrollment.
Time Frame: 12 months post-drug product infusion through Month 24
Population: TP included all participant who received beti-cel.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
g/dL | 10.653 (1.5096)

13. Secondary Outcome: Unsupported Total Hb Levels at Month 6, 9, 12, 18 and 24
Description: Unsupported total Hb level was defined as the total Hb measurement level without any acute or chronic pRBC transfusions within 60 days prior to the measurement date.
Time Frame: At Month 6, 9, 12, 18 and 24
Population: TP included all participant who received beti-cel. Here, "overall number of participants analyzed" signifies those participants who had a least 1 unsupported total Hb measurement during Study HGB-212 and "number analyzed" signifies those participants who had an unsupported total Hb measurement at the specific timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 17
g/dL
  At Month 6 | 10.41 (1.253)
  At Month 9 | 10.61 (1.338)
  At Month 12 | 10.65 (1.619)
  At Month 18: number analyzed (Participants) | 15
  At Month 18 | 11.00 (1.483)
  At Month 24 | 10.82 (1.580)

14. Secondary Outcome: Number of Participants With Unsupported Total Hb Levels (>=10 g/dL, >=11 g/dL, >=12 g/dL, >=13 g/dL, and >=14 g/dL) at Months 6, 9, 12, 18 and 24
Description: Number of participants with unsupported total Hb levels (>=10 g/dL, >=11 g/dL, >=12 g/dL, >=13 g/dL, and >=14 g/dL) meeting the thresholds were reported at Months 6, 9, 12, 18 and 24. Participants were evaluable if they had an unsupported total Hb measurement at the specific timepoint, where unsupported total Hb level is defined as the total Hb measurement level without any acute or chronic pRBC transfusions within 60 days prior to the measurement date.
Time Frame: At Months 6, 9, 12, 18 and 24
Population: TP included all participants who received beti-cel. Here, "Overall number of participants analyzed" signifies those participants who had a least 1 unsupported total Hb measurement during Study HGB-212 and "number analyzed" signifies those participants who had an unsupported total Hb measurement at the specific timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 17
Participants
  At Month 6 (>=10 g/dL) | 11
  At Month 6 (>=11 g/dL) | 4
  At Month 6 (>=12 g/dL) | 3
  At Month 6 (>=13 g/dL) | 1
  At Month 6 (>=14 g/dL) | 0
  At Month 9 (>=10 g/dL) | 13
  At Month 9 (>=11 g/dL) | 5
  At Month 9 (>=12 g/dL) | 3
  At Month 9 (>=13 g/dL) | 1
  At Month 9 (>=14 g/dL) | 0
  At Month 12 (>=10 g/dL) | 12
  At Month 12 (>=11 g/dL) | 6
  At Month 12 (>=12 g/dL) | 3
  At Month 12 (>=13 g/dL) | 2
  At Month 12 (>=14 g/dL) | 1
  At Month 18 (>=10 g/dL): number analyzed (Participants) | 15
  At Month 18 (>=10 g/dL) | 13
  At Month 18 (>=11 g/dL): number analyzed (Participants) | 15
  At Month 18 (>=11 g/dL) | 5
  At Month 18 (>=12 g/dL): number analyzed (Participants) | 15
  At Month 18 (>=12 g/dL) | 3
  At Month 18 (>=13 g/dL): number analyzed (Participants) | 15
  At Month 18 (>=13 g/dL) | 3
  At Month 18 (>=14 g/dL): number analyzed (Participants) | 15
  At Month 18 (>=14 g/dL) | 0
  At Month 24 (>=10 g/dL) | 10
  At Month 24 (>=11 g/dL) | 7
  At Month 24 (>=12 g/dL) | 3
  At Month 24 (>=13 g/dL) | 3
  At Month 24 (>=14 g/dL) | 1

15. Secondary Outcome: Percentage of Participants Who Have Not Received Chelation Therapy for At Least 6 Months Following Drug Product Infusion
Description: Percentage of participants who have not received chelation therapy for at least 6 months following drug product infusion were reported.
Time Frame: From 6 to 24 months
Population: TP included all participant who received beti-cel.
Measure: Number; unit: Percentage of participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
Percentage of participants | 61.1

16. Secondary Outcome: Time From Last Iron Chelation Use to Last Follow-up
Description: Time from last iron chelation use to last follow-up to 24 months was reported.
Time Frame: From last Iron Chelation up to Month 24 (actual maximum time frame of up to approximately 29 months due to visit window)
Population: TP included all participants who received beti-cel. Participants were evaluable for this endpoint if they had not received iron chelation therapy for at least 6 months following drug product infusion. Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome. Data are presented through the Month 24 Visit based on calendar dates and including visit windows.
Measure: Median (Full Range); unit: Months
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 13
Months | 17.81 [0.3 to 28.9]

17. Secondary Outcome: Number of Participants Who Used Therapeutic Phlebotomy Post Drug Product Infusion
Description: Therapeutic phlebotomy could be used in lieu of chelation in participants who had Hb consistently >= 11 g/dL and who were no longer receiving regular transfusions, at the discretion of the investigator. Number of participants who used therapeutic phlebotomy post Drug Product infusion for up to Month 24 were reported.
Time Frame: From drug product infusion through Month 24
Population: TP included all participants who received beti-cel.
Measure: Count of Participants; unit: Participants
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
Participants | 2

18. Secondary Outcome: Annualized Phlebotomy Therapy Usage Following Drug Product Infusion
Description: Annualized phlebotomy therapy usage (number of procedures per year, calculated from DP infusion through last follow-up) were reported.
Time Frame: From drug product infusion through Month 24
Population: TP included all participants who received beti-cel. Here, "Overall number of participants analyzed" signifies those participants who received therapeutic phlebotomy.
Measure: Mean (Standard Deviation); unit: Number of procedures per year
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 2
Number of procedures per year | 4.22 (3.192)

19. Secondary Outcome: Change From Baseline in Liver Iron Content by Magnetic Resonance Imaging (MRI)
Description: Change From Baseline in Liver Iron Content by MRI at Months 12 and 24 were reported. Baseline is defined as value closest to but prior to conditioning.
Time Frame: Baseline, Month 12 and 24
Population: TP included all participants who received beti-cel. Participants were evaluable for TI if they had completed the study (i.e., completed the Month 24 Visit), achieved TI, or did not achieve TI during the study. Here, "number analyzed" signifies those participants who had LIC data available at Baseline, Months 12 and 24.
Measure: Mean (Standard Deviation); unit: milligram per gram (mg/g)
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
milligram per gram (mg/g)
  Change at Month 12: number analyzed (Participants) | 17
  Change at Month 12 | 3.171 (5.4134)
  Change at Month 24 | 1.033 (4.4407)

20. Secondary Outcome: Change From Baseline in Cardiac T2* on MRI
Description: Change From Baseline in Cardiac T2* on MRI from Baseline, Month 12 and 24 was reported.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Participants were evaluable for TI if they had completed the study (i.e., completed the Month 24 Visit), achieved TI, or did not achieve TI during the study. Here, "number analyzed" signifies those participants who were evaluable at specific timepoint.
Measure: Median (Full Range); unit: milliseconds
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
milliseconds
  Change at Month 12: number analyzed (Participants) | 17
  Change at Month 12 | -0.2 [-27 to 7]
  Change at Month 24 | 0.2 [-33 to 12]

21. Secondary Outcome: Change From Baseline in Serum Ferritin
Description: Serum ferritin was commonly used for an indirect estimation of body iron stores. Although sensitive, it is not specific for iron overload as it can be elevated in a variety of infectious and inflammatory states, and in the presence of cytolysis. Change from baseline in serum ferritin at Months 12 and 24 was reported.
Time Frame: Baseline, Month 12 and 24
Population: TP included all participants who received beti-cel. Participants are evaluable for TI if they had completed the study (i.e., completed the Month 24 Visit), achieved TI, or did not achieve TI during the study. Here, "number analyzed" signifies those participants who were evaluable at specific timepoint.
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 18
picomole per liter (pmol/L)
  Change at Month 12: number analyzed (Participants) | 17
  Change at Month 12 | 87.3 (1302.76)
  Change at Month 24 | -605.2 (1716.90)

22. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL) Total Scores at Months 12 and 24
Description: PedsQL GCS designed to measure health-related quality of life in pediatric and adolescents (2-18 years). It encompassed 4 dimensions of functioning (physical [8 items], emotional [5 items], social [5 items], school [3 items]). Age groups: Toddler (2-4 years), Young pediatric (5-7 years), Pediatric (8-12 years), Teens (13-18 years). The questionnaire was also completed by parent/caregiver to assess parents' perceptions of their children's quality of life. The Toddler group consisted of 21 items, using a 5-point Likert scale (0 to 4); all other groups consisted of 23 items, with a 3-point Likert scale (0, 2, 4) for young pediatric, a 5-point Likert scale for pediatric and teens groups. All reported scores were transformed on a scale from 0 to 100 for each domain where 0=100, 1=75, 2=50, 3=25, and 4=0. Higher scores correspond with higher quality of life.
Time Frame: Baseline, Month 12 and 24
Population: TP included all participants who received beti-cel. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome and "number analyzed" signifies those participants who were evaluable at specific timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 13
Score on a scale
  Parent total score: Change at Month 12 | -6.20 (12.948)
  Parent total score: Change at Month 24: number analyzed (Participants) | 12
  Parent total score: Change at Month 24 | -3.49 (19.621)
  Patient total score: Change at Month 12: number analyzed (Participants) | 11
  Patient total score: Change at Month 12 | 2.96 (14.857)
  Patient total score: Change at Month 24: number analyzed (Participants) | 11
  Patient total score: Change at Month 24 | 4.84 (11.321)

23. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension Youth Scale (EQ-5D-Y) VAS Health Status at Months 12 and 24
Description: EQ-5D is a validated, standardized, generic instrument that was most widely used preference based health related quality of life questionnaire in cost effectiveness and health technologies assessment. EQ-5D-Y was a version of instrument specifically developed and validated for use by youths aged 12 through 17 years. The EQ-5D-Y visual analog scale (VAS) consisted of a 20-cm vertical VAS, with anchors of 0 (worst imaginable health state) and 100 (best imaginable health state). Respondents were asked to rate their own health state today by drawing a line from a box containing these words to the point on the scale that they felt most accurately reflected their current health state. The VAS was reported (raw data) on a scale of 0-100 where 0= death and 100= perfect health. Higher scores corresponded with higher quality of life.
Time Frame: Baseline, Months 12 and 24
Population: TP included all participants who received beti-cel. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 7
Score on a scale
  Health State: Change at Month 12 | 0.3 (11.91)
  Health State: Change at Month 24 | 2.0 (12.33)

24. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension Adult Scale (EQ-5D-3L) VAS Heath Status Score at Months 12 and 24
Description: EQ-5D is a validated, standardized, generic instrument that was most widely used preference based health related quality of life (HRQoL) questionnaire in cost effectiveness and health technologies assessment. Participants age >=18 at time of informed consent were eligible to complete the EQ-5D-3L visual analog scale (VAS) which consisted of a 20-cm vertical VAS, with anchors of 0 (worst imaginable health state) and 100 (best imaginable health state). Respondents were asked to rate their own health state today by drawing a line from a box containing these words to the point on the scale that they felt most accurately reflected their current health state. The VAS was reported (raw data) on a scale of 0-100 where 0= death and 100= perfect health. Negative change in score indicated decrease in quality of life (as measured by EQ5D VAS) from baseline.
Time Frame: Baseline, Months 12 and 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 5
Score on a scale
  Health State: Change at Month 12 | -3.6 (13.13)
  Health State: Change at Month 24 | -2.4 (10.50)

25. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) Questionnaire Total Score
Description: FACT-BMT is assessed bone marrow transplant related quality of life in adults. Total score was sum of sub-scale scores for 5 domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and Bone Marrow Transplantation Subscale. Each item scored on a 5-point Likert scale based on participant agreement with each statement: 0 for "not at all," 1 for "a little bit," 2 for "somewhat," 3 for "quite a bit," and 4 for "very much. Reported scores were transformed as follows: After taking into account reverse scores for questions constructed in negative form, subscale score for each domain was calculated by multiplying sum of item scores by number of items in subscale, then dividing by number of items answered. Total score was sum of subscale total added together and ranges from 0-148. Higher scores corresponded with higher quality of life.
Time Frame: Baseline, Months 12 and 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 4
Score on a scale
  Total Score: Change at Month 12 | 0.33 (6.716)
  Total Score: Change at Month 24 | 2.58 (4.246)

26. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36), Version 2, Acute (Physical and Mental Component Summary Scores) at Months 12 and 24
Description: SF-36 was designed to measure health-related quality of life in adults. The instrument consisted of 36 items that were aggregated into 8 multi-item scales (physical functioning [1=yes, limited a lot, to 3=no, not limited at all], role-physical [1=all of time, to 5=none of time], bodily pain [1=very severe, to 6=none], general health [1=poor, to 5=excellent], vitality [1=none of time, to 5=all of time], social functioning [1=all of time, to 5=none of time], role emotional [1=all of time, to 5=none of time] and mental health [1=all of time, to 5=none of the time]). The 8 scales were summarized as Physical Component Summary (PCS) score (physical functioning, role-physical, bodily pain, general health scales) and Mental Component Summary (MCS) score (vitality, social functioning, role-emotional, mental health scales). Reported summary scores were transformed on a scale from 0-100 (higher scores corresponded with higher quality of life), with change from baseline results being presented.
Time Frame: Baseline, Months 12 and 24
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | LentiGlobin BB305 Drug Product
Number analyzed (Participants) | 5
Score on a scale
  Physical Component Summary: Change at Month 12 | -0.89 (10.289)
  Physical Component Summary: Change at Month 24 | 1.09 (8.167)
  Mental Component Summary: Change at Month 12 | 2.42 (7.637)
  Mental Component Summary: Change at Month 24 | 2.08 (7.281)

ADVERSE EVENTS:
Time Frame: From date of informed consent to the date of last followup (an average of 32.5 months of followup for ITT subjects).
Description: ITT population included all participants who initiated any study procedures, beginning with mobilization by G-CSF and/or plerixafor.
Arm/Group | LentiGlobin BB305 Drug Product
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 6/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LentiGlobin BB305 Drug Product (N=19)
Cardiac failure congestive (Cardiac disorders) | 1
Headache (Nervous system disorders) | 1
Pyrexia (General disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1
Soft tissue infection (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LentiGlobin BB305 Drug Product (N=19)
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 1
Adverse drug reaction (General disorders) | 1
Application site pain (General disorders) | 1
Application site swelling (General disorders) | 1
Catheter site pain (General disorders) | 4
Fatigue (General disorders) | 3
Feeling cold (General disorders) | 1
Injection site reaction (General disorders) | 1
Mucosal inflammation (General disorders) | 7
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 3
Puncture site pain (General disorders) | 2
Pyrexia (General disorders) | 7
Hypersensitivity (Immune system disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 2
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 3
Blood creatinine increased (Investigations) | 1
Blood testosterone decreased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Coombs direct test positive (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Pulmonary function test decreased (Investigations) | 1
Transaminases increased (Investigations) | 2
Weight decreased (Investigations) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Post procedural discomfort (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 9
Skin abrasion (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ageusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 11
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 16
Neutrophilia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Ear pain (Ear and labyrinth disorders) | 1
Chalazion (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 3
Anal inflammation (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Oral pain (Gastrointestinal disorders) | 1
Palatal ulcer (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 12
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic mass (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 12
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Delayed puberty (Endocrine disorders) | 1
Hypogonadism (Endocrine disorders) | 1
Secondary hypogonadism (Endocrine disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Bronchitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 3
Cystitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lice infestation (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 3
Pyelonephritis (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Systemic infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Varicella zoster virus infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 2
Vulvovaginal candidiasis (Infections and infestations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Hyperchloraemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Vitamin K deficiency (Metabolism and nutrition disorders) | 1

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of participants analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT03207009/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03207009/SAP_001.pdf